CLINICAL TRIAL: NCT06174285
Title: Effect of Psychedelic VR-augmented Therapy on Patients With Clinical Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tartu (Other)
Collaborators: Confido Medical Centre (Unknown)
Responsible Party: Principal Investigator, Karl Kristjan Kaup, Junior Research Fellow, University of Tartu
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DB-RCT-PSYRREAL
Record Dates: First submitted 2023-11-22; First posted 2023-12-18 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psyrreal (Experimental): Psychedelic virtual reality experience.
  Interventions: Other: Therapeutic Intervention with Psychedelic Virtual Reality
- Routine Realms (Sham Comparator): A non-psychedelic virtual reality experience that is largely analogous to Psyrreal.
  Interventions: Other: Therapeutic Intervention with Non-Psychedelic Virtual Reality
- No intervention (No Intervention): A conditional waiting list condition. This condition may be included, dependent on the availability of sufficient participants and resources.

INTERVENTIONS:
Other: Therapeutic Intervention with Psychedelic Virtual Reality — A 55-minute immersive psychedelic virtual reality experience is incorporated into a therapeutic intervention, comprising a preparatory phase and a subsequent integration session based on the individual's experience.
  Arms: Psyrreal
Other: Therapeutic Intervention with Non-Psychedelic Virtual Reality — A 55-minute immersive virtual reality experience is incorporated into a therapeutic intervention, comprising a preparatory phase and a subsequent integration session based on the individual's experience.
  Arms: Routine Realms

SUMMARY:
Research has demonstrated that psychedelic compounds possess significant therapeutic potential for a variety of disorders, including depression. Despite these findings, the underlying mechanisms driving the therapeutic efficacy of psychedelics remain elusive. Furthermore, there exists a debate over the contribution of the subjective psychedelic experience to their therapeutic benefits. In this study, virtual reality (VR) is utilized as a tool to replicate the subjective experiences induced by psychedelics, aiming to explore their impact on depressive symptoms within a clinical sample.

The primary objective of this research is to examine the influence of psychedelic-like phenomenology, as simulated through VR, on depressive symptoms. The study is structured into two distinct arms: the experimental condition features 'Psyrreal,' a VR experience designed to emulate psychedelic effects and the control condition which includes 'Routine Realms,' an analogous VR experience devoid of psychedelic elements. A third waiting list condition may be included, dependent on the availability of sufficient participants and resources. Additionally, the study seeks to identify and analyze various potential mediators that might underpin the therapeutic outcomes observed.

ELIGIBILITY:
Inclusion Criteria:

* Persistent depressive symptoms observed during the initial screening and confirmed at baseline, as determined through a comprehensive psychiatric evaluation.
* Provision of written informed consent by the participant.
* Fluent in Estonian as a native language.

Exclusion Criteria:

* Presence of significant impairments in vision, hearing, or balance.
* Active suicidal ideation or current engagement in self-harm behaviors. Note: Individuals meeting this criterion will be directed to suitable crisis intervention services.
* Established diagnosis of bipolar disorder.
* Manifestation of psychotic symptoms.
* History of schizophrenia, either personally or within two generations of the family lineage.
* Ongoing diagnosis of epilepsy, dementia, or any other neurological condition that could interfere with the effective utilization of virtual reality (VR) technology.
* Susceptibility to motion sickness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Emotional State Questionnaire 2 depression subscale score from baseline to follow-up | Measured at 3 time-points - on the day 1 of intervention, and two weeks and two months after intervention.
  Measurement of the intensity of depressive symptoms during a specified period (suitable for periods longer than a week).

SECONDARY OUTCOMES:
Short mood questionnaire | Measured at two time-points - baseline and on the day 1 of the intervention..
  A short questionnaire based on the Emotional State Questionnaire 2 to evaluate changes in mood on a short time-scale.
Emotional State Questionnaire 2 other subscales | Measured at 3 time-points - on the day 1 of intervention and two weeks and two months after intervention.
  These subscales measure symptoms of panic disorder, agoraphobia, generalized anxiety disorder, asthenia and sleeping disorder.
State Mindfulness Scale | Measured at two time-points -baseline and on the day 1 of the intervention
  Questionnaire for evaluating change in state mindfulness due to virtual reality experience.
Adapted short version of the questionnaire for the assessment of altered states of consciousness (11D-ASC) | Measured at one time-point - after the virtual reality experience on the day 1 of the intervention.
  Questionnaire to evaluate alterations in consciousness during the virtual reality experience. Some items are adapted for implementation in virtual reality and a subset of questions are omitted from the original 11D-ASC questionnaire.
Psychological Insight Questionnaire | Measured at one time-point - after the virtual reality experience on the day 1 of the intervention.
  Questionnaire for measuring psychological insight during acute (psychedelic) experiences.
Ego-Dissolution Inventory | Measured at one time-point - after the virtual reality experience on the day 1 of the intervention.
  Questionnaire for measuring the experience of ego-dissolution during the virtual reality experience.
Avoidance/Acceptance-Promoting Experience Questionnaire | Measured at one time-point - after the virtual reality experience on the day 1 of the intervention.
  Questionnaire for measuring changes in acceptance- and avoidance-related beliefs due to virtual reality experiences.
Awe Experience Scale | Measured at one time-point - after the virtual reality experience on the day 1 of the intervention.
  Questionnaire for measuring the experience of awe during the virtual reality experience.

OTHER OUTCOMES:
Custom background questionnaire part I | Measured at one time-point - before the virtual reality experience on the day 1 of the intervention.
  Contains items regarding demographic information and prior experiences with virtual reality.
Custom background questionnaire part II | Measured at one time-point - at the two month follow-up.
  Contains items on prior experiences with psychedelics and spiritual practices, and the subjective impression of the intervention.
Semi-structured interview transcriptions | Measured at one time-point - immediately after the virtual reality experience on the day 1 of the intervention.
  If the participant agrees, the post-experience integration session will be recorded and transcribed.

CONTACTS AND LOCATIONS:
Overall Officials: Jaan Aru, PhD, Principal Investigator — University of Tartu
Locations (1):
- Confido Medical Centre, Tallinn, Harju, Estonia